CLINICAL TRIAL: NCT02941328
Title: A Phase II, Mono-center, Placebo-controlled, Double-blind, Crossover Trial to Investigate Effect and Efficacy of Pyridostigmine in Dutch Patients With Spinal Muscular Atrophy Types 2, 3 and 4
Brief Title: SPACE Trial: Pyridostigmine vs Placebo in SMA Types 2, 3 and 4
Acronym: SPACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Camiel Wijngaarde, MD, UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL38048.041.14
Record Dates: First submitted 2016-09-30; First posted 2016-10-21 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Spinal Muscular Atrophy; SMA; Kugelberg-Welander Disease
Keywords: SMA, SMN1, Kugelberg-Welander
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood; Spinal Muscular Atrophy, Type IV | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pyridostigmine (Experimental): (this is a cross-over trial, in which participants will receive both a placebo and pyridostigmine in different study periods. Both investigators and participants are blinded for what medication is used in what period. All patients will eventually use a placebo for 8 weeks and pyridostigmine for 8 weeks).
  Interventions: Drug: Pyridostigmine
- Placebo (Placebo Comparator): (this is a cross-over trial, in which participants will receive both a placebo and pyridostigmine in different study periods. Both investigators and participants are blinded for what medication is used in what period. All patients will eventually use a placebo for 8 weeks and pyridostigmine for 8 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyridostigmine — Pyridostigmine, administered orally starting with 2mg/kg/day (in 4 daily doses, i.e. 0,5mg/kg/dose) and slowly increasing to a maximum dosage of 6mg/kg/day (4 daily doses of 1,5mg/kg/day)
  Other Names: Mestinon
  Arms: Pyridostigmine
Drug: Placebo — Placebo administered orally starting with 2mg/kg/day (in 4 daily doses, i.e. 0,5mg/kg/dose) and slowly increasing to a maximum dosage of 6mg/kg/day (4 daily doses of 1,5mg/kg/day)
  Arms: Placebo

SUMMARY:
A trial investigating the effects of pyridostigmine (mestinon) versus a placebo in a double-blind cross over trial in patients with hereditary proximal spinal muscular atrophy (SMA) types 2, 3 and 4.

DETAILED DESCRIPTION:
In this cross-over trial we will investigate the effects of pyridostigmine (mestinon) versus a placebo on fatigability in patients with hereditary proximal spinal muscular atrophy (SMA) types 2, 3 and 4 (aged 12 and older) The study participants will be using a placebo during 8 weeks and mestinon during 8 weeks. Both investigators and patients are blinded to the treatment allocation in both periods. Patients will be randomly assigned to use placebo or mestinon first. At the end of the study, patients will have used both mestinon and a placebo during 8 weeks.

In both phases (periods) of the cross over study, study medication dosage will slowly be increased to a maximum dosage of 6 mg/kg/day (spread over 4 doses daily) in order to either prevent side effects or to manage them as good as possible. This scheme allows us to assist our participants in case side effects do occur early. Although we strive to have all patients on the same dosage per kg of body weight, serious side effects will obviously lead to lowering the dosage.

Before the start of medication use (either placebo or pyridostigmine), baseline measurements will be taken: a physical examination and data concerning both primary and secondary outcomes (MFM, MRC scores, fatigability tests, etc.) will be collected. After use a drug (mestinon/placebo) for 8 weeks these tests will be repeated, to evaluate possible medication effect. After a wash-out period of approximately 1-2 weeks the same scheme is used for the second study period (i.e. the cross-over design). Unblinding follows after the entire study is completed (i.e.: last included patients finishes participation).

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of SMA type 2, 3a, 3b or 4
* Genetically confirmed homozygous SMN1 deletion
* Ability to complete visits during trial period;
* Given oral and written informed consent when ≥18 years old;
* Given informed consent by the parents or legal representative(s) in case of patients aged ≥12 till <18 years old (in accordance with Dutch law)
* Ability of performing at least 2 subsequent rounds of the Nine Hole Peg test
* A maximum total Motor Function Measure (MFM) score of 80% (i.e.: a maximum score under 80% of the D1+D2+D3 subscores).

Exclusion Criteria:

* Known concomitant disorders of the NMJ (e.g. but not limited to: Lambert Eaton myasthenic syndrome, myasthenia gravis);
* Use of drugs that may alter NMJ function
* Classic SMA type 1;
* Apprehension against participation in EMG;
* Inability to meet study visits;
* Mechanical gastro-intestinal, urinary or biliary obstruction;
* Clinical significant alterations of laboratory tests (electrolytes, liver function, kidney function, thyroid function or blood dysplasia) drawn within 14 days prior to start of study entry;
* ECG abnormalities known as a contraindication for pyridostigmine use;
* Current pregnancy or breast-feeding
* Allergy to bromides
* Severe bronchial asthma (in case of uncertainty of diagnosis, we will contact treating pulmonologist or physician)
* Total MFM score at baseline (screening) > 80% (i.e.: a maximum total MFM score above 80% of the D1+D2+D3 subscores).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
MFM (Motor Function Measurement). | change over the course of 8 weeks compared to baseline
  D1+D2+D3 but also D1, D2, or D3 sub scores of the MFM scales will be used.
repeated nine-hole peg test performance | Change in performance (in time to complete) the test rounds over the course of 8 weeks of medication compared to baseline
  The time needed tot complete multiple rounds of the nine hole peg test (hence: repeated NHPT) will be recorded (visit 1) and compared to the performance on the test after 8 weeks of treatment (placebo or mestinon) (visit 2). Visit 3 will serve as the baseline measurement for the 2nd study period (again followed by 8 weeks of treatment and the final study visit (visit 4)).

SECONDARY OUTCOMES:
endurance nine hole peg test | Change in performance after 8 weeks of therapy (placebo or mestinon).
  During the endurance tests, patients will perform at 75% of their maximum performance. Differences in before and after treatment results (number of rounds completed) will be analysed
endurance box-and-block test | Change in performance after 8 weeks of therapy (placebo or mestinon)
  During the endurance tests, patients will perform at 75% of their maximum performance. Differences in before and after treatment results (number of rounds completed) will be analysed. This test will be performed only if the patient is capable of performing it.
endurance walk test | Change in performance after 8 weeks of therapy (placebo or mestinon).
  During the endurance tests, patients will perform at 75% of their maximum performance. Differences in before and after treatment results (e.d. total distance travelled) will be analysed. This test will be performed only if the patient is able to walk.

CONTACTS AND LOCATIONS:
Overall Officials: W.L. Van der Pol, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center of Utrecht (UMCU), Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stam M, Wijngaarde CA, Bartels B, Asselman FL, Otto LAM, Habets LE, van Eijk RPA, Middelkoop BM, Goedee HS, de Groot JF, Roes KCB, Schoenmakers MAGC, Nieuwenhuis EES, Cuppen I, van den Berg LH, Wadman RI, van der Pol WL. Randomized double-blind placebo-controlled crossover trial with pyridostigmine in spinal muscular atrophy types 2-4. Brain Commun. 2022 Dec 9;5(1):fcac324. doi: 10.1093/braincomms/fcac324. eCollection 2023. PMID 36632180
- [Derived] Stam M, Wadman RI, Wijngaarde CA, Bartels B, Asselman FL, Otto LAM, Goedee HS, Habets LE, de Groot JF, Schoenmakers MAGC, Cuppen I, van den Berg LH, van der Pol WL. Protocol for a phase II, monocentre, double-blind, placebo-controlled, cross-over trial to assess efficacy of pyridostigmine in patients with spinal muscular atrophy types 2-4 (SPACE trial). BMJ Open. 2018 Jul 30;8(7):e019932. doi: 10.1136/bmjopen-2017-019932. PMID 30061431